CLINICAL TRIAL: NCT03082508
Title: A Pivotal Trial to Establish the Efficacy and Safety of Algisyl in Patients With Moderate to Severe Heart Failure
Acronym: AUGMENT-HFII
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: LoneStar Heart, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LSH-14-001
Record Dates: First submitted 2017-03-13; First posted 2017-03-17 (Actual); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Heart Failure; Dilated Cardiomyopathy; Heart Failure With Reduced Ejection Fraction
Keywords: Algisyl; Heart Failure; Dilated Cardiomyopathy; Alginate Hydrogel; Heart Failure with Reduced Ejection Fraction; Congestive Heart Failure
MeSH Terms: conditions — Heart Failure; Cardiomyopathy, Dilated | interventions — Drug Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Algisyl (Experimental): Algisyl device (implants) administered during a surgical procedure.
  Interventions: Device: Algisyl
- Standard Medical Therapy (Active Comparator): as per protocol
  Interventions: Drug: Standard Medical Therapy

INTERVENTIONS:
Device: Algisyl — Algisyl device (implants) administered during a surgical procedure
  Other Names: intramyocardial injections of alginate hydrogel
  Arms: Algisyl
Drug: Standard Medical Therapy — as per protocol
  Other Names: Evidence based therapy for heart failure; heart failure medications; drug therapy
  Arms: Standard Medical Therapy

SUMMARY:
AUGMENT-HF II is a study to evaluate the efficacy and safety of the Algisyl device. The purpose of this study is to investigate Algisyl employed as a method of left ventricular augmentation and restoration in patients with dilated cardiomyopathy.

Algisyl will be injected into the myocardium under direct visualization during the surgical procedure. Structural abnormalities in the heart are known to play a central role in HF, and clinical evidence supports a strong causal relationship between cardiac chamber dilation and heart failure. Because dilation, and not contractile dysfunction, appears to be responsible for the severity of the disease, the mitigation or prevention of the deleterious structural abnormalities of the left ventricle appears to be an important therapeutic target for patients with this life threatening illness.

Hence, a therapy that specifically reduces LV wall stress, targets LV dilatation and LV remodeling may offer an important new alternative in the treatment of heart failure. Algisyl is being investigated based on evidence that suggests an ability of the implants to reduce wall stress, reshape the LV chamber and reduce the LV chamber size as well as prevent the progressive ventricular dilation and remodeling associated with HF.

The physiologic response to progressive exercise using direct measures of ventilation and gas exchange via the cardiopulmonary exercise test is an important diagnostic tool in the management of the patient with HF, quantifying responses to therapy, and as a reliable prognostic utility for predicting outcomes in patients with HF.

Numerous studies have established the strong association of peak VO2 with mortality and morbidity risk in HF. Peak VO2 conceptually is considered an overall global marker of cardiopulmonary health and is a reflection of the degree of impairment in ventricular function ( the heart's pumping capacity), oxygen delivery and oxygen utilization.

Hence, employing the change in peak VO2 as a primary endpoint in this clinical study provides a strong objective measure that can be interpreted in independent blinded fashion, to evaluate the result of the therapeutic intervention and provide an equally strong assessment of the prognostic implications for patients in the study.

This clinical evaluation is intended to provide confirmatory evidence of the effectiveness and safety of the device Algisyl in patients with advanced heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. The patients must be able and willing to give written informed consent
2. The patients will be adult (age ≥ 18 years and ≤ 79 years) males or females
3. The patients must be on stable, evidence-based therapy for heart failure

   Evidence-based therapy for heart failure is defined as an ACE-inhibitor (ACE-I), and/or angiotensin II receptor blockers (ARB) for patients at stable doses for 1 month prior to enrollment, if tolerated, and a beta blocker (carvedilol, metoprolol succinate, Nebivolol or bisoprolol) for 3 months prior to enrollment, if tolerated. Recent up-titration of the beta blocker is acceptable if the patient has been stable on this dose for 1 month prior to enrollment. Stable is defined as no more than a 100% increase or a 50% decrease in dose. Contraindications or intolerance to therapies should be documented. In those intolerant to both ACE-I and ARB, combination therapy with hydralazine and oral nitrate should be considered. Therapeutic equivalence for ACE-I substitutions is allowed within the enrollment stability timelines. Aldosterone inhibitor therapy should be added when NYHA Class III or IV symptoms occur on standard therapy. If aldosterone inhibitor therapy is to be administered in NYHA Class II patients, it must be initiated and optimized prior to enrollment. Eplerenone requires dosage stability for 1 month prior to enrollment. Diuretics should be used as necessary to keep the patient euvolemic. All heart failure therapeutics and dosages should be documented in the Case Report Forms.
4. The patient must have cardiac resynchronization therapy (CRT) if clinically indicated, implanted ≥3 months prior to randomization.

   * Note: In those patients not receiving CRT or CRT-D therapy the investigator should not anticipate initiating this therapy within 6 months after randomization
5. The patient must have an implanted cardio-defibrillator (ICD) if clinically indicated, implanted at least 30 days prior to randomization.

   *Note: If the patient has clinical indications for an ICD but refuses the ICD, this refusal of ICD therapy must be document in the medical record and the patient may be enrolled with this documentation.
6. The patients will have a left ventricular ejection fraction equal to or less than 35% via echocardiography, cardiac catheterization, radionuclide scan, or magnetic resonance imaging (measured within the last 30 days)
7. The patients will have a left ventricular end diastolic dimension indexed to body surface area (LVEDDi) of greater than or equal to 30 mm/m2 (LVEDD/BSA) and an LVEDD of greater than or equal to 85 mm (measured within the last 30 days)
8. Patients must have symptomatic heart failure with a Peak VO2 of 9.0 - 15.0 ml/min/kg (performed using a treadmill). Patients must perform two CPX tests (within 30 days of randomization and performed at least 20 hours apart) that differ by no more than 15% in the observed value for Peak VO2 and have a mean value of 9.0 - 15.0 ml/min/kg from these two tests. All CPX tests performed for the study must have a Peak Respiratory Exchange Ratio (RER) of at least 1.0 to be accepted as a valid test.
9. Patient's surgical risk must be considered reasonable and the evaluation of surgical risk should include review of coronary and left ventricular angiography. Surgical risk assessment should include the consideration of risk presented by prior surgical procedures such as prior mid-sternotomy surgical procedures.

   *Note: investigators should observe standard clinical practice for the management of antithrombotic therapy in patients undergoing surgical procedures in accordance with the American College of Chest Physicians Guidelines: Perioperative management of antithrombotic therapy: Antithrombotic Therapy and Prevention of Thrombosis, 9th edition
10. If female, the patients must be (a) post-menopausal, (b) surgically sterile, or (c) using adequate birth control and have a negative serum pregnancy test within 7 days prior to administration of study device

Exclusion Criteria:

1. Patients for whom it is planned to receive CABG, MVR, heart transplantation or LVAD within the next 6 months.
2. Patients presenting with cardiogenic shock.
3. Patients presenting with a restrictive cardiomyopathy such as due to amyloidosis, sarcoidosis, or hemochromatosis
4. Patient with a history of constrictive pericarditis
5. Patients with a Q wave myocardial infarction (MI) within the last 30 days
6. Patients with a recent history of stroke (within 60 days prior to the surgical procedure)
7. A left ventricular (LV) wall thickness of the LV free-wall, at the mid-ventricular level, of less than 8 mm (screening echocardiography must confirm a minimum wall thickness of 8 mm)
8. Patients with an estimated glomerular filtration rate (GFR) < 30 mL/min/1.73 m2
9. Clinically significant liver enzyme abnormalities, i.e., AST(SGOT) and ALT (SGPT) more than 2.5 times the upper limit of normal
10. History of severe COPD (i.e., FEV 1< 1 liter or FEV1 < 50% predicted)
11. The patients will not be receiving concurrently an Investigational Product in another clinical trial or have received an investigational Product in another clinical trial in the 30 days prior to enrollment
12. A life expectancy of less than 1 year or any other condition that, in the opinion of the clinical investigator, might compromise any aspect of the trial

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Peak VO2 | 6 months
  Change in Peak VO2 from baseline to 6 months of follow-up
Primary Safety Endpoint: Death or Re-hospitalization for Worsening Heart Failure | 12 months
  Death or Re-hospitalization for Worsening Heart Failure

SECONDARY OUTCOMES:
NYHA Functional Class | 6 months
  NYHA Functional Class
Six-minute walk distance | 6 months
  Six minute walk distance
Peak VO2 at 12 months | 12 months
  Change in Peak VO2 from baseline to 12 months of follow-up
QOL | 6 months
  Quality of Life as measured by KCCQ (Kansas City Cardiomyopathy Questionnaire)

OTHER OUTCOMES:
MACE-free survival | 30 days, 6 months, 12 months
  Major Adverse Cardiovascular Events (MACE)-free survival at 30 days, 6 months and 12 months
MACE | 30 days, 6 months, 12 months
  Occurrence of individual MACE components at 30 days, 6 months and 12 months
MAE | 30 days, 6 months, 12 months
  Major Adverse Events at 30 days, 6 months and 12 months
Afib | 30 days, 6 months, 12 months
  Overall incidence of atrial fibrillation and freedom from atrial fibrillation

IPD SHARING:
Plan to Share IPD: No